CLINICAL TRIAL: NCT01355783
Title: A Phase 3 Trial of E7777 in Combination With CHOP Compared With CHOP Alone for the First-Line Treatment of Peripheral T-cell Lymphoma
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E7777-G000-301
Record Dates: First submitted 2011-05-16; First posted 2011-05-18 (Estimated); Last update posted 2013-11-18 (Estimated); Status verified 2013-11

CONDITIONS: Peripheral T-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — E7777 fusion protein

ARMS (2):
- E7777 + CHOP Chemotherapy (Active Comparator)
  Interventions: Drug: E7777
- CHOP alone (Active Comparator)
  Interventions: Drug: E7777

INTERVENTIONS:
Drug: E7777 — Treatment in both arms is for 6 cycles at 21 days/cycle.

SUMMARY:
The purpose of this study is to evaluate whether treatment of E7777 in combination with CHOP has superior efficacy compared with CHOP alone in improving complete response rate (CRR) in first line treatment of subjects with Peripheral T-cell Lymphoma (PTCL).

ELIGIBILITY:
Inclusion:

Subjects must meet all of the following criteria to be included in the study:

1. Local pathologic diagnosis of PTCL with the following histology types: PTCL, not otherwise specified (PTCL-NOS), angioimmunoblastic T-cell lymphoma (AITL), and anaplastic large cell lymphoma (ALCL) (ALK-negative or ALKpositive with IPI ≥ 2).
2. Stage II, III or IV disease.
3. Tumor lesion(s) measurable in 2 dimensions by computed tomography (CT) and is at least 20 mm in the longest transverse dimension for non-lymph node masses and at least 20 mm in longest transverse dimension for lymph nodes. Subcutaneous masses can be used as indicator lesions. If the lesion was previously irradiated, it must have progressed prior to randomization (by investigator assessment) to be used as a measurable lesion.
4. Tumor biopsy available for central pathologic review; may be archived sample from prior biopsy within 6 months of study enrollment, or sample to be obtained on study during screening.
5. Age ≥ 18 years.
6. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
7. Adequate bone marrow reserve as evidenced by:

   * absolute neutrophil count (ANC) ≥ 1000/mm3 (1.0x109/L)
   * platelets ≥ 50,000/mm3 (50x109/L); (≥ 25,000/mm3 [25x109/L] allowed if thrombocytopenia secondary to bone marrow involvement by lymphoma)
   * hemoglobin ≥ 8 g/dL (80 g/L)
8. Adequate liver function as evidenced by:

   * bilirubin ≤ 1.5 times the upper limit of normal (ULN)
   * aspartate aminotransferase (AST [SGOT]) and alanine aminotransferase (ALT [SGPT]) ≤ 3 times the ULN (≤ 5 times the ULN if hepatic involvement)
   * albumin ≥ 3.0 g/dL (30 g/L)
9. Adequate renal function as evidenced by serum creatinine ≤ 2.0 mg/dL (176 μmol/L) or calculated creatinine clearance ≥ 40 mL/min per the Cockcroft-Gault formula.
10. Willing and able to comply with all aspects of the protocol.
11. Written informed consent prior to any study-specific screening procedures.
12. Female subjects of childbearing potential must have a negative serum betahuman chorionic gonadotropin (β-hCG) pregnancy test at Screening and a negative serum or urine β-hCG pregnancy test result at Baseline, and must agree to use a highly effective method of contraception (see protocol for list) throughout the entire study period and for 30 days after study drug discontinuation.
13. Male subjects who are partners of women of childbearing potential must use or their partners must use a highly effective method of contraception (see protocol for list) beginning at least 1 menstrual cycle prior to starting study drug(s),throughout the entire study period, and for 30 days after study drug discontinuation, unless they are sexually abstinent or have undergone a successful vasectomy. Those with partners using hormonal contraceptives must also be using an additional approved method of contraception, as described previously.

Exclusion:

Subjects who meet any of the following criteria will be excluded from the study:

1. Diagnosis of ALCL ALK-positive with IPI 0 or 1, adult T-cell leukemia/lymphoma (ATLL), precursor T-cell lymphoblastic lymphoma/leukemia, extranodal NK/TCL nasal type, enteropathy-associated TCL, hepatosplenic TCL, subcutaneous panniculitis-like TCL, and cutaneous T-cell lymphoma (CTCL) including mycosis fungoides and Sezary syndrome.
2. Known central nervous system (CNS) involvement with lymphoma.
3. Prior chemotherapy, immunotherapy, denileukin diftitox, or investigational agent(s) for this lymphoma, with the exception that a single cycle of CHOP (or CHOP-based therapy) is allowed if the last dose of CHOP (or CHOP-based therapy) was administered ≤ 28 days before study enrollment (Lead-In) or randomization (Main Study).
4. Prior radiotherapy for this lymphoma, with the following exception: prior radiation therapy for localized disease ≥ 4 weeks before randomization is allowed as long as the irradiated area is not at the mediastinal area or at the site of the only potentially measurable disease.
5. Prior malignancy within past 5 years (except non-melanoma skin cancer or carcinoma in situ of the cervix).
6. Serious intercurrent illness.
7. Significant cardiac disease requiring ongoing treatment, including congestive heart failure (CHF), severe coronary artery disease (CAD), cardiomyopathy, uncontrolled cardiac arrhythmia, unstable angina pectoris, or myocardial infarction (MI) (within 6 months of study enrollment).
8. Left ventricular ejection fraction (LVEF) less than institutional lower limit of normal, as determined by multigated acquisition scan (MUGA) or echocardiogram.
9. Major surgery within 2 weeks of study enrollment.
10. Active infections requiring specific anti-infective therapy.
11. Known human immunodeficiency virus (HIV) infection; known active hepatitis B or hepatitis C infection.
12. Deep vein thrombosis within 3 months of study enrollment.
13. Females who are pregnant (positive urine test) or breastfeeding.
14. Any history of or concomitant medical condition that, in the opinion of the Investigator, would compromise the subject's ability to safely complete the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-03; Primary Completion 2014-10 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
To evaluate whether treatment of E7777 in combination with CHOP chemotherapy has superior efficacy compared with CHOP alone in improving progression-free survival (PFS) in first line treatment of subjects with peripheral T-cell lymphoma | pre-randomization 4 weeks until disease progression
  * Pretreatment or pre-randomization (screening and baseline): 4 weeks.
  * Treatment: 18 weeks.
  * Follow up: 2 to 3 years after the end of study treatment. Treatment will stop upon disease progression, unacceptable toxicity, or death, whichever occurs first. The Investigator or subject may also stop study treatment at any time for safety or personal reasons; however subject should remain on study, if possible, for follow-up.

SECONDARY OUTCOMES:
To evaluate whether E7777 in combination with CHOP treatment has superior efficacy compared with CHOP treatment alone as assessed by overall survival (OS) and by transplant rate.· To compare safety of E7777 in combination with CHOP | pre-randomization 4 weeks until disease progression
  * Pretreatment or pre-randomization (screening and baseline): 4 weeks.
  * Treatment: 18 weeks.
  * Follow up: 2 to 3 years after the end of study treatment. Treatment will stop upon disease progression, unacceptable toxicity, or death, whichever occurs first. The Investigator or subject may also stop study treatment at any time for safety or personal reasons; however subject should remain on study, if possible, for follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Chean Eng Ooi, Study Director — Eisai Inc.
Locations (2):
- United States (2):
  - Skokie, Illinois
  - Morristown, New Jersey